CLINICAL TRIAL: NCT07314788
Title: Empathy and Virtual Reality (VR)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jennifer Britton, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20241195
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Virtual Reality; Fear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fear-inducing Virtual Reality (VR) experience (Experimental): Participants will complete a single virtual reality (VR) exposure lasting approximately 1-2 minutes, involving a fear-inducing scenario (e.g., walking a plank above a high-rise building or canyon).
  Interventions: Behavioral: Fear-inducing Virtual Reality (VR) experience
- Neutral Virtual Reality (VR) experience (Active Comparator): Participants will complete a single virtual reality (VR) exposure lasting approximately 1-2 minutes, involving a neutral scenario (e.g., walking to the edge of a curb at street level).
  Interventions: Behavioral: Neutral Virtual Reality (VR) experience

INTERVENTIONS:
Behavioral: Fear-inducing Virtual Reality (VR) experience — Participants will complete a single virtual reality (VR) exposure involving a fear-inducing scenario (e.g., walking a plank above a high-rise building or canyon).
  Arms: Fear-inducing Virtual Reality (VR) experience
Behavioral: Neutral Virtual Reality (VR) experience — Participants will complete a single virtual reality (VR) exposure involving a fear-inducing scenario (e.g., walking to the edge of a curb at street level).
  Arms: Neutral Virtual Reality (VR) experience

SUMMARY:
This study will characterize the subjective and physiological changes associated with empathy following a fear-inducing virtual reality (VR) experience.

ELIGIBILITY:
Inclusion Criteria:

* College-aged adults (18-25 years old)
* English-speaking
* Normal or corrected vision.
* Able to provide consent.

Exclusion Criteria:

• Presence of a significant and/or unstable medical illness (e.g., cardiovascular disease, cancer, neurological disorder) or head trauma (e.g., concussion).

Additional exclusion criteria apply to virtual reality (VR):

* VR contraindications: epilepsy, migraines, flu, sleep deprivation, etc.
* More than minimal VR experience assessed via self-report (e.g., How often have you used virtual reality in the past? 0=never, 6=very frequently)
* Extreme phobia of heights and/or spiders will be assessed using Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) specific phobia subscale.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported empathy scores | Baseline (prior to VR experience) and approximately 5 minutes post-VR experience.
  Participant will view videos of other individuals undergoing a fear-inducing virtual reality (VR) experience and will self-report level of empathy on a scale 0=not at all to 10=extremely. Average empathy ratings will be compared pre-VR and post-VR.
Change in heart rate | Baseline (prior to VR experience) and approximately 5 minutes post-VR experience.
  Average heart rate (beats/minute) will be collected while watching videos of other individuals undergoing a fear-inducing virtual reality (VR) experience and will be compared pre-VR and post-VR.

SECONDARY OUTCOMES:
Change in the correlation between self-reported anxiety scores of self and another | Baseline (prior to VR experience) and approximately 5 minutes post-VR experience.
  Participant will view videos of other individuals undergoing a fear-inducing virtual reality (VR) experience and will self-report level of anxiety on self and other on a scale 0=not at all, 10=extremely. Anxiety ratings of self and another will be correlated and compared pre-VR and post-VR. Greater correlation will reflect greater alignment of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Britton, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No